CLINICAL TRIAL: NCT04719429
Title: The Effects of Dietary Protein Source on Postprandial Plasma Amino Acid Availability, Gut-derived Appetite Regulating Hormones, and Subjective Appetite Sensations in Young Males
Brief Title: The Effects of Cricket- and Beef-derived Protein on Plasma Amino Acid Concentrations and Appetite Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Tyler A. Churchward-Venne, Ph.D., Assistant Professor, McGill University, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A08-M28-18B
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Aminoacidemia; Appetitive Behavior
Keywords: dietary protein; insect protein; young men; beef collagen; amino acids; appetite
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricket-derived protein beverage (Experimental): Ingestion of a cricket-derived protein beverage
  Interventions: Dietary Supplement: Cricket-derived Protein
- Beef-derived protein beverage (Experimental): Ingestion of a beef-derived protein beverage
  Interventions: Dietary Supplement: Beef-derived Protein

INTERVENTIONS:
Dietary Supplement: Cricket-derived Protein — Beverage containing 25 g cricket-derived protein
  Arms: Cricket-derived protein beverage
Dietary Supplement: Beef-derived Protein — Beverage containing 25 g beef-derived protein
  Arms: Beef-derived protein beverage

SUMMARY:
Dietary protein plays an important role in appetite regulation. Source of ingested dietary protein may have different effects on appetite, satiety, and/or food intake in humans. Insects are a rich source of protein consumed by many people around the world; however, the capacity of insect-derived protein to regulate appetite and food intake is unclear. The purpose of this study was to compare postprandial plasma glucose, insulin, amino acid, and appetite regulatory hormone concentrations, subjective appetite sensations, and food intake following the ingestion of 25 g of cricket- and beef-derived protein in healthy young males.

DETAILED DESCRIPTION:
With the rapid increase in the global population, the production of sufficient amounts of conventional animal-based protein to meet global dietary demands may no longer be desired nor feasible. Insects may represent an environmentally sustainable additional source of dietary protein that has the potential to help ensure global food security in the future. However, the functional characteristics of insect-derived proteins when fed to humans is unclear. Further, how insect-derived proteins compare to other animal-derived proteins (e.g. from beef) have not been explored.

The purpose of this study was to compare postprandial plasma glucose, insulin, and amino acid concentrations, gut-derived appetite regulatory hormones, subjective appetite sensations, and ad libitum energy intake following the ingestion of 25 g insect- or beef-derived protein in healthy young men. It was hypothesized that hyperaminoacidaemia would be more rapid following the ingestion of beef-derived protein compared to cricket-derived protein, although total amino acid availability would be similar between protein sources over a 300-minute postprandial period. It was further hypothesized there would be no difference between protein sources on postprandial subjective appetite sensations or subsequent ad libitum energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18-35 years inclusive
* Healthy, moderately active
* BMI < 30 kg/m2 and > 18.5 kg/m2
* Having given informed consent

Exclusion Criteria:

* Presence of any identified metabolic or intestinal disorders
* Use of tobacco products
* Adherence to a strict vegetarian or vegan diet
* Use of medications known to affect protein metabolism
* Allergy to shellfish or crustaceans
* Allergy to beef protein
* Engagement in physical exercise training more than 6 days per week

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Plasma leucine concentration | 0-5 hours in the post-prandial period
  umol/L
Subjective appetite sensations (hunger, fullness, desire to eat, prospective food consumption) | 0-5 hours in the post-prandial period
  mm (visual analogue scale)

SECONDARY OUTCOMES:
Plasma branched-chain amino acid concentration | 0-5 hours in the post-prandial period
  umol/L
Plasma essential amino acid concentration | 0-5 hours in the post-prandial period
  umol/L
Plasma non-essential amino acid concentration | 0-5 hours in the post-prandial period
  umol/L
Plasma total amino acid concentration | 0-5 hours in the post-prandial period
  umol/L
Plasma glucose | 0-5 hours in the post-prandial period
  mmol/L
Plasma insulin | 0-5 hours in the post-prandial period
  pmol/L
Plasma GLP-1 | 0-5 hours in the post-prandial period
  pg/mL
Plasma PYY | 0-5 hours in the post-prandial period
  pg/mL
Ad libitum food energy intake | assessed 5 hours after protein intake
  kJ

CONTACTS AND LOCATIONS:
Overall Officials: Tyler A Churchward-Venne, Ph.D., Principal Investigator — McGill University
Locations (1):
- Exercise Metabolism and Nutrition Research Laboratory, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No